CLINICAL TRIAL: NCT02164097
Title: A Pilot Study to Evaluate the Safety and Preliminary Evidence of an Effect of ODSH (2-O, 3-O Desulfated Heparin) in Accelerating Platelet Recovery in Pediatric Patients With a Recurrent Solid Tumor Receiving "ICE" Chemotherapy
Brief Title: ODSH + ICE Chemotherapy in Pediatric Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYMC-165
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Recurrent Solid Tumor; Refractory Solid Tumor; Sarcoma; Wilms' Tumor; Neuroblastoma
Keywords: ICE; ODSH; platelet recovery; recurrent solid tumor
MeSH Terms: conditions — Sarcoma; Wilms Tumor; Neuroblastoma | interventions — N-desulfated,2-O,3-O-desulfated heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ODSH and ICE Chemotherapy (Experimental): Patients will receive standard doses of ICE Chemotherapy:
  * Ifosfamide 1800 mg/m2 mixed with Mesna 360 mg/m2 IV over 2 hours on days 1, 2, 3, 4, and 5
  * Carboplatin 400 mg/m2 IV over 1 hour on days 1 and 2
  * Etoposide 100 mg/m2 IV over 1 hour on days 1, 2, 3, 4, and 5
  ODSH will be administered as a 4 mg/kg bolus 30 minutes after the first ifosfamide dose followed immediately by a continuous intravenous ODSH infusion of 0.25 mg/kg/hour for five consecutive days, on days 1-5, for a total of 120 hours of continuous ODSH infusion.
  Interventions: Drug: ODSH

INTERVENTIONS:
Drug: ODSH
  Other Names: 2-O, 3-O Desulfated Heparin

SUMMARY:
This study will be with pediatric patients who have refractory/recurrent solid tumors. They will receive standard chemotherapy (ICE) and we are investigating if the addition of a new drug, ODSH, will help to increase the time of their platelet recovery after ICE chemotherapy.The purpose of this study is to evaluate the safety and tolerability of ODSH in pediatric patients receiving "ICE" chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or refractory solid tumors. This may include, but is not limited to, osteosarcoma, chondrosarcoma, Ewing's sarcoma, Wilm's Tumor, medulloblastoma, neuroblastoma, hepatoblastoma, rhabdomyosarcoma, retinoblastoma, and primitive neuroectodermal tumors. Histologic proof malignancy must have been available at the time of initial diagnosis.
* Age: 1-21
* Patients must have received standard first-line chemotherapy or other appropriate standard first line therapy for their malignancy.
* Patients must have radiologic or histologic evidence of recurrence
* Patients must have fully recovered from the toxic effects of the prior chemotherapy and must have an ANC >1000/μL and a platelet count >100,000/μL
* Performance status > 60 from Lansky (age 1 to 16) or Karnofsky (age > 16)
* Adequate hepatic and renal function (AST, ALT, bilirubin and creatinine < 2.5 x upper normal limit).
* Parent or guardian able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Patients who, in the investigator's opinion, have extensive bone marrow involvement with tumor
* Presence of significant active infection or uncontrolled bleeding
* Renal insufficiency, which, in the opinion of the investigator, might adversely affect schedule and dose of therapy ICE chemotherapy. patients with creatinine levels ≥2 mg/dl are not eligible
* Pre-existing liver disease , other than liver metastasis
* Use of recreational drugs within the prior month
* Known history of positive hepatitis B surface antigens or HCV antibodies
* Known history of positive test for HIV antibodies
* Patients receiving any form of anticoagulant therapy
* Presence of a known bleeding disorder or coagulation abnormality
* Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to study entry
* Pregnant or breast-feeding patients
* Patient with childbearing potential not using adequate contraception
* Hemorrhage risk that requires maintenance of platelet counts at 50,000 or higher.
* Psychiatric or neurologic conditions that could compromise patient safety or compliance, or interfere with the ability of the patient or family to give proper informed consent.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine if ODSH is safe in pediatric patients | 60 days following last dose of ODSH
  All patients will be followed for 60 days after the last dose of ODSH in a treatment cycle in which ODSH is administered. All serious adverse events related to ODSH will be monitored.

SECONDARY OUTCOMES:
To see if ODSH has a positive effect on platelet recovery | 60 days after last dose of ODSH
  Platelet counts will be monitored to determine when the platelet count remained > 100,000 after nadir for two consecutive days in the absence of a prior platelet transfusion within the previous 48 hours in pediatric patients receiving "ICE" chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States